CLINICAL TRIAL: NCT02255058
Title: Psychometric Validation of the Multi-INdependency Dimensions (MIND) Score for Patients Under Prolonged Mechanical Ventilation
Brief Title: MIND Score for Prolonged Mechanical Ventilation
Acronym: MIND
Status: Completed | Type: Observational
Sponsor: Linde AG (Industry)
Responsible Party: Sponsor
Other Study IDs: Linde001
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2014-10

CONDITIONS: Functional Test, COPD, Neuromuscular Disorders, Mechanical Ventilation, Weaning, Disability
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — The study is a Prospective observational cohort study

SUMMARY:
It was decided to develop a comprehensive disability score specifically designed for patients receiving prolonged mechanical ventilation (PMV); the collection of information included in the score should not impose any further intervention beyond what is routinely performed. So a new questionnaire was created (called the Multi-INdependency Dimensions (MIND) that included 3 sections (nurse, physiotherapist and medical doctor), 11 categories and 18 items. Each question was adapted to have a 5 item Likert scale.

The primary objective of the study will be to evaluate the psychometric performance of the MIND score in terms of validity, reliability and sensitivity to change over time. The secondary objective will be to assess the inclusion of biological markers on the overall performance of the MIND score

DETAILED DESCRIPTION:
Following recruitment all participants will be assessed by a medical doctor or respiratory therapist (trained on the study) who will fill out the MIND questionnaire on admission and make sure the other scales/questionnaires are also completed. On the same day of the collection of MIND, MRC score for quadriceps and biceps strength, Sequential Organ Failure Assessment (SOFA) score, Glasgow coma scale, Hospital Anxiety-depression scale (HADS), EuroQol-5D, Gussago Dependence Nursing Scale (GNS) will be also gathered. After 1 day and 30 days the MIND questionnaire will be also evaluated. Index of ADL-(Katz index) will be evaluated on discharge as well as weaning rate and survival.

Sample Size Determination

Based on the method of Rouquette A et al (1) we estimated a sample size of 200 patients to allow for the Rasch modelling to be applied.

Statistical analysis

Assessment of construct validity:

Confirmation of the structure (e.g. multitrait analysis), clinical validity (comparison of disability score according to external clinical criteria)

Assessment of reliability:

Internal consistency reliability (using Cronbach's alpha), test-retest reliability (using intraclass correlations)

Assessment of sensitivity to change over time:

Comparison of change in disability score according to change in external clinical criteria Guidance for interpretation of disability score: Estimation of thresholds for patients' classification

1-Rouquette A, Falissard B Sample size requirements for the internal validation of psychiatric scales Int J Methods Psychiatr Res. 2011 Dec;20(4):235-49. doi: 10.1002/mpr.352. Epub 2011 Oct 24.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Prolonged mechanical Ventilation and a Diagnosis of Acute lung injury, COPD/Chronic Lung Disease, Neuromuscular Disorders, Post-Operative, Cardiovascular Disorders, Trauma, Other.

Exclusion Criteria:

* Expected length of stay <48h, unable to achieve consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Prolonged mechanical Ventilation and a Diagnosis of Acute lung injury, COPD/Chronic Lung Disease, Neuromuscular Disorders, Post-Operative, Cardiovascular Disorders, Trauma, Other.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the psychometric performance of the MIND score in terms of validity, reliability and sensitivity to change over time | 6 Months

SECONDARY OUTCOMES:
To assess the inclusion of biological markers on the overall performance of the MIND score | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Joao C Winck, MD,PhD, Study Director — Linde AG, Global Business Unit Healthcare
Locations (5):
- REMEO El Pilar, Buenos Aires, Argentina
- Colombia (2):
  - REMEO Bogota, Bogotá
  - REMEO Medellin, Medellín
- Germany (2):
  - REMEO Centre, Berlin
  - REMEO Mahlow, Berlin

REFERENCES:
- [Derived] Winck JC, Gilet H, Kalin P, Murcia J, Plano F, Regnault A, Dreher M, Vitacca M, Ambrosino N. Validation of the Multi-INdependence Dimensions (MIND) questionnaire for prolonged mechanically ventilated subjects. BMC Pulm Med. 2019 Jun 20;19(1):109. doi: 10.1186/s12890-019-0870-2. PMID 31221129